CLINICAL TRIAL: NCT06244329
Title: The Application of Repetitive Transcranial Magnetic Stimulation (rTMS) as an Adjunct Therapy in Reduction of Craving and Consumption of Illicit Drugs
Brief Title: Repetitive Transcranial Magnetic Stimulation in Drugs Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20210602002
Record Dates: First submitted 2024-01-27; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-10

CONDITIONS: Substance Use Disorders
Keywords: Transcranial Magnetic Stimulation; Substance Use Disorders; Craving
MeSH Terms: conditions — Substance-Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A blinded assessor, who is not aware of the condition order, conducts all behavioral assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High frequency repetitive transcranial magnetic stimulation (Experimental): 10 Hz rTMS is applied to the left dorsolateral prefrontal cortex (DLPFC). The individual DLPFC is located using the Beam F3 method. The stimulation intensity is 100% of the resting motor threshold of the left primary motor cortex. Each session of stimulation lasts for around 9 mins. We apply 6-session rTMS, with 2-3 times per week.
  Interventions: Device: Transcranial magnetic stimulation
- Sham repetitive transcranial magnetic stimulation (Experimental): Sham rTMS is applied to the left dorsolateral prefrontal cortex (DLPFC). The individual DLPFC is located using the Beam F3 method. The stimulation intensity is 20% of the resting motor threshold of the left primary motor cortex, which is deemed completely ineffective in modulating brain excitability. We apply 6-session sham rTMS, with 2-3 times per week.
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Transcranial Magnetic Stimulation (TMS) uses magnetic fields to stimulate nerve cells in the brain. TMS uses a small electromagnetic coil controlled by a computer program to deliver short, powerful pulses of magnetic energy focused precisely on parts of the brain's pre-frontal cortex. High-frequency repetitive TMS can enhance the excitability of the stimulated region.

SUMMARY:
This study also aims to develop and apply a standard repetitive transcranial magnetic stimulation (rTMS) protocol on drug users. The investigators want to focus on the effects of rTMS on amphetamine and cocaine as they are the most commonly used types of illicit drugs in Hong Kong.

The primary research question is:

• To examine if rTMS can reduce craving and consumption of the most commonly used illicit drugs (amphetamine, cocaine) among people with drug use disorders in Hong Kong?

The secondary research questions are:

* What is the association between rTMS protocol (frequency, intensity) and drug craving and consumption?
* Would there be gains in executing functioning among participants who have received rTMS treatment?
* Would there be a reduction in depressive and anxiety symptoms among participants who have received rTMS treatment?

The investigators would use a cross-over design (figure 1) to investigate the effects of rTMS. The investigators would recruit participants through community drug rehabilitation and youth outreach services. Participants who meet the selection and exclusion criteria will be invited to join. Upon obtaining their written consent, the investigators would randomize participants to a treatment (rTMS) group and a sham stimulation (placebo) group. Upon completing the first phase (2 weeks), there would be a washout period of 2 weeks. The two groups will swap (treatment becomes sham, and vice-versa) and the second phase will proceed. A double-blinded procedure will be implemented. Outcome measures will be conducted at baseline, after Phase I, at the start of Phase II, and at the end of Phase II.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 60.
2. Illicit drug users in the community (not in institutions).
3. Uses either amphetamine (ice) and/or cocaine frequently (at least 4 times per week).
4. Craving Visual Analogue Scale (VAS, 11-point from 0 - 10) score of at least 5 or above on either amphetamine or cocaine.
5. Interest in participating in drug treatment or rehabilitation or have already engaged in such services offered by health or social services.
6. Not engaged in pharmacological or physical treatment related to substance use disorders in past six months.

Exclusion Criteria:

1. Have a history of seizures or a family history of epilepsy.
2. Have severe mental disorders like bipolar disorder or psychosis.
3. Have brain damage from illness or injury, such as a brain tumor, a stroke or a traumatic brain injury.
4. Have any metal or implanted medical devices in the body.
5. Have frequent or severe headaches.
6. Pregnant or thinking of becoming pregnant.
7. Had prior treatment with rTMS in the past year.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Craving | Baseline (before the phase I intervention)
  An 11-item Craving Experience Questionnaire (CEQ), a theory-based and concise assessment tool for measuring substance cravings, is utilized. Each item is rated on a scale of 0 to 10, resulting in a total score range of 0 to 110. A higher score indicates a higher level of craving.
Craving | 3-week post intervention (after 6-session of the phase I intervention)
  An 11-item Craving Experience Questionnaire (CEQ), a theory-based and concise assessment tool for measuring substance cravings, is utilized. Each item is rated on a scale of 0 to 10, resulting in a total score range of 0 to 110. A higher score indicates a higher level of craving.
Craving | Baseline (before the phase II intervention)
  An 11-item Craving Experience Questionnaire (CEQ), a theory-based and concise assessment tool for measuring substance cravings, is utilized. Each item is rated on a scale of 0 to 10, resulting in a total score range of 0 to 110. A higher score indicates a higher level of craving.
Craving | 3-week post intervention (after 6-session of the phase II intervention)
  An 11-item Craving Experience Questionnaire (CEQ), a theory-based and concise assessment tool for measuring substance cravings, is utilized. Each item is rated on a scale of 0 to 10, resulting in a total score range of 0 to 110. A higher score indicates a higher level of craving.

SECONDARY OUTCOMES:
Readiness for change | Baseline (before the phase I intervention)
  The Contemplation Ladder which measures the motivation for change, is used. The motivation for change is rated on a scale of 0 (No thought about quitting. I cannot live without drugs) to 10 (I have changed my drug use and will never go back to the way I used drugs before), with a total score of 10. A higher score means a higher motivation for change.
Readiness for change | 3-week post intervention (after 6-session of the phase I intervention)
  The Contemplation Ladder which measures the motivation for change, is used. The motivation for change is rated on a scale of 0 (No thought about quitting. I cannot live without drugs) to 10 (I have changed my drug use and will never go back to the way I used drugs before), with a total score of 10. A higher score means a higher motivation for change.
Readiness for change | Baseline (before the phase II intervention)
  The Contemplation Ladder which measures the motivation for change, is used. The motivation for change is rated on a scale of 0 (No thought about quitting. I cannot live without drugs) to 10 (I have changed my drug use and will never go back to the way I used drugs before), with a total score of 10. A higher score means a higher motivation for change.
Readiness for change | 3-week post intervention (after 6-session of the phase II intervention)
  The Contemplation Ladder which measures the motivation for change, is used. The motivation for change is rated on a scale of 0 (No thought about quitting. I cannot live without drugs) to 10 (I have changed my drug use and will never go back to the way I used drugs before), with a total score of 10. A higher score means a higher motivation for change.
Drug Consumption | Baseline (before the phase I intervention)
  A self-report questionnaire Set 6 of Beat Drug Fund (BDF)-Hong Kong, which assesses drug use frequency in past two weeks, is used. The patients are required to indicate their usage of each type of drug by selecting one of the following options: Never used, Used occasionally, and Used regularly.
Drug Consumption | 3-week post intervention (after 6-session of the phase I intervention)
  A self-report questionnaire Set 6 of Beat Drug Fund (BDF)-Hong Kong, which assesses drug use frequency in past two weeks, is used. The patients are required to indicate their usage of each type of drug by selecting one of the following options: Never used, Used occasionally, and Used regularly.
Drug Consumption | Baseline (before the phase II intervention)
  A self-report questionnaire Set 6 of Beat Drug Fund (BDF)-Hong Kong, which assesses drug use frequency in past two weeks, is used. The patients are required to indicate their usage of each type of drug by selecting one of the following options: Never used, Used occasionally, and Used regularly.
Drug Consumption | 3-week post intervention (after 6-session of the phase II intervention)
  A self-report questionnaire Set 6 of Beat Drug Fund (BDF)-Hong Kong, which assesses drug use frequency in past two weeks, is used. The patients are required to indicate their usage of each type of drug by selecting one of the following options: Never used, Used occasionally, and Used regularly.
Trail Making Test | Baseline (before the phase I intervention)
  A test of speed of processing
Trail Making Test | 3-week post intervention (after 6-session of the phase I intervention)
  A test of speed of processing
Trail Making Test | Baseline (before the phase II intervention)
  A test of speed of processing
Trail Making Test | 3-week post intervention (after 6-session of the phase II intervention)
  A test of speed of processing
Continuous Performance Test-Identical Pairs (CPT-IP) | Baseline (before the phase I intervention)
  A computer-administered measure of sustained attention
Continuous Performance Test-Identical Pairs (CPT-IP) | 3-week post intervention (after 6-session of the phase I intervention)
  A computer-administered measure of sustained attention
Continuous Performance Test-Identical Pairs (CPT-IP) | Baseline (before the phase II intervention)
  A computer-administered measure of sustained attention
Continuous Performance Test-Identical Pairs (CPT-IP) | 3-week post intervention (after 6-session of the phase II intervention)
  A computer-administered measure of sustained attention
Mazes test from The Neuropsychological Assessment Battery® (NAB®) | Baseline (before the phase I intervention)
  Mazes test is used to measure reasoning and problem-solving.
Mazes test from The Neuropsychological Assessment Battery® (NAB®) | 3-week post intervention (after 6-session of the phase I intervention)
  Mazes test is used to measure reasoning and problem-solving.
Mazes test from The Neuropsychological Assessment Battery® (NAB®) | Baseline (before the phase II intervention)
  Mazes test is used to measure reasoning and problem-solving.
Mazes test from The Neuropsychological Assessment Battery® (NAB®) | 3-week post intervention (after 6-session of the phase II intervention)
  Mazes test is used to measure reasoning and problem-solving.
The Depression Anxiety Stress Scale (DASS)-short form | Baseline (before the phase I intervention)
  The anxiety and depression subscales (13 items) of DASS is used for monitoring the negative emotional states of the participants. The total score is 39 with a higher scores indicating a higher level of emotional problems.
The Depression Anxiety Stress Scale (DASS)-short form | 3-week post intervention (after 6-session of the phase I intervention)
  The anxiety and depression subscales (13 items) of DASS is used for monitoring the negative emotional states of the participants. The total score is 39 with a higher scores indicating a higher level of emotional problems.
The Depression Anxiety Stress Scale (DASS)-short form | Baseline (before the phase II intervention)
  The anxiety and depression subscales (13 items) of DASS is used for monitoring the negative emotional states of the participants. The total score is 39 with a higher scores indicating a higher level of emotional problems.
The Depression Anxiety Stress Scale (DASS)-short form | 3-week post intervention (after 6-session of the phase II intervention)
  The anxiety and depression subscales (13 items) of DASS is used for monitoring the negative emotional states of the participants. The total score is 39 with a higher scores indicating a higher level of emotional problems.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No